CLINICAL TRIAL: NCT03092154
Title: Lipid-lowering Agents in Patients With Dermatomyositis and Polymyositis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Samuel Katsuyuki Shinjo, PhD, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MYO-HCFMUSP-03
Record Dates: First submitted 2017-03-09; First posted 2017-03-27 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Treatment Side Effects
MeSH Terms: interventions — Hypolipidemic Agents; Therapeutics

STUDY DESIGN:
Intervention Model Description: Two groups: with or without lipid-lowering agents
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposed (Experimental): Patients will receive lipid-lowering agents (Artovastatin) for at least 12-weeks
  Interventions: Drug: Lipid-lowering agents (Artovastatin)
- No intervention (No Intervention): Patients will not receive artovastatin (lipid-lowering agents)

INTERVENTIONS:
Drug: Lipid-lowering agents (Artovastatin) — Artovastatin 20 mg /day, orally, 12 consecutive weeks.
  Other Names: Therapy
  Arms: Exposed

SUMMARY:
The use of lipid lowering agents in patients with idiopathic inflammatory myopathies is controversial. Therefore, the aim of the present study is to assess clinically and laboratory the impact of lipid-lowering agents in this population.

DETAILED DESCRIPTION:
Impact of the lipid lowering agents on patients with dermatomyositis and polymyositis.

ELIGIBILITY:
Inclusion Criteria:

* fullfill all criteria of Bohan and Peter (1975)
* dyslipidemia
* age> 18 years
* prednisone ≤ 0.25 mg/kg/day (or ≤ 15mg/ ay) in the last three months
* without changing nutritional habits in the last three months, and during the study period
* no change of lifestyle in the last three months, and during the study period

Exclusion Criteria:

Patients with:

* disease relapsing
* overlapping myositis
* neoplasia associated myositis
* diabetes mellitus
* current and/or chronic infections
* patients undergoing major surgery within six months prior to the study
* pregnant patients
* previous use of lipid-lowering agents in the last 6 months
* in the use of cyclosporin, erythromycin, clarithromycin, fibrates, niacin, azole antifungals, cimetidine, diltiazem
* active liver disease or persistent elevations of hepatic enzymes, with no apparent cause, exceeding three times the upper limit of normality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Endothelial function | 12 weeks
  Ultrasound-based measurements of brachial reactivity were performed according to the guidelines of the International Brachial Artery Reactivity Task Force. The assessment of vascular reactivity was carried out by the same examiner. The left brachial artery was measured at a longitudinal section above the antecubital fossa, using a high-resolution ultrasound system Sequoia Echocardiography System, version 6.0, Acuson; Siemens, Vernon, CA) equipped with a multifrequency linear transducer (7-12 MHz) to produce two-dimensional images. This technique was used to evaluate the change in arterial diameter and blood flow after physical and pharmacological stimulation.

SECONDARY OUTCOMES:
Side effects | 12 weeks
  Side effects of lipid-lowering agents
Patient/Parent Global Activity | 12 weeks
  This partially validated tool measures the global evaluation by the patient, or by the parent if the patient is a minor, of the patient's overall disease activity at the time of assessment using a 10 cm. visual analogue scale.
Physician Global Activity | 12 weeks
  This partially validated tool measures the global evaluation by the treating physician of the overall disease activity of the patient at the time of assessment using a 10 cm. visual analogue scale and a 5 point Likert scale.
Manual Muscle Testing | 12 weeks
  This partially validated tool assesses muscle strength using manual muscle testing (MMT). A 0 - 10 point scale is proposed for use. An abbreviated group of 8 proximal, distal, and axial muscles performs similarly to a total of 24 muscle groups, and is also proposed for use for research studies.
Muscle enzymes | 12 weeks
  This partially validated tool measures the serum activities of at least 2 of the 4 muscle-associated enzymes including creatine phosphokinase (CK), the transaminases (ALT, AST), lactate dehydrogenase (LD) and aldolase.
Myositis Disease Activity Assessment Tool | 12 weeks
  After local anesthesia, a cutaneous incision will be made in lateral thigh face. The biopsy will be done using the Bergstrom needle. Histological (hematoxylin and eosin)/immunohistochemical (CD4, CD8, CD68, CD20, C5b-9, MHCI, MHCII, CD31) analysis will be performed in muscle samples (at baseline and after 12 weeks) in all patients (present study)
Health Assessment Questionnaire | 12 weeks
  Especific questionnaire (health assessment questionnaire). Pontuaction 0.00-3.00

CONTACTS AND LOCATIONS:
Overall Officials: Samuel K Shinjo, PhD, Principal Investigator — Universidade de Sao Paulo - Rheumatology Division
Locations (1):
- Samuel Katsuyuki Shinjo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No